CLINICAL TRIAL: NCT02670304
Title: The Randomized Controlled Trial Study of Letrozole in the Prevention of Medium and Severe Ovarian Hyperstimulation Syndrome in Invitro Fertilization Treatment
Brief Title: Preventive Application of Letrozole Decrease Incidence of Early Onset of OHSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhou Canquan, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 28843020
Record Dates: First submitted 2013-08-07; First posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: letrozole; ovarian hyperstimulating syndrome
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Letrozole; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- letrozole (Experimental): letrozole for the first day after ovum picked up at least for 5 days.
  Interventions: Drug: letrozole
- aspirin (Active Comparator): asprin for the first day after ovum picked up at least for 5 days.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: letrozole — letrozole from the day of oocyte retrieval for 5 days
  Other Names: Femara
  Arms: letrozole
Drug: Aspirin — aspirin from the day of oocyte retrieval for 5 days
  Arms: aspirin

SUMMARY:
Letrozole is one kind of aromatase inhibitors which may have effect on decrease estrogen in luteal phase and inhibit the luteal function of ovary. In 2009, Letrozole was reported as one candidate for the treatment or prevention of ovarian hyperstimulation syndrome.

DETAILED DESCRIPTION:
Letrozole was proved to be effective in decreasing the estradiol level of luteal phase after ovum picked up. In this randomized controlled study, investigators try to observe the effectiveness of letrozole on decreasing the incidence of early ovarian hyperstimulation syndrome and vascular epithelium growth factor level of women with high ovarian hyperstimulation syndrome risks.

ELIGIBILITY:
Inclusion Criteria:

* infertile women undergoing IVF treatment with more than 25 oocytes collected.

Exclusion Criteria:

* letrozole contraindications,e.g. severe hepatic and renal dysfunction

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
incidence of early OHSS | up to 1 months

SECONDARY OUTCOMES:
vascular endothelial growth factor level | up to 1 months
  vascular endothelial growth factor in pg/ml
incidence of hydrothorax | up to 1 months
incidence of liver dysfunction | up to 1 months
incidence of renal dysfunction | up to 1 months
incidence of electrolytic imbalance | up to 1 months
incidence of hemoconcentration | up to 1 months
incidence of elevated WBC | up to 1 months

IPD SHARING:
Plan to Share IPD: No
no plan to make IPD available